CLINICAL TRIAL: NCT06506929
Title: The Effect of Task Specific Physical Therapy for Persons With Advanced Multiple Sclerosis
Brief Title: Task Specific Training for Advanced Multiple Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: Multiple Sclerosis Foundation (Unknown)
Responsible Party: Principal Investigator, Herb Karpatkin, Associate professor, Hunter College of City University of New York
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0303
Record Dates: First submitted 2024-07-03; First posted 2024-07-18 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Pilot study- single group pretest postest
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Task specific Physical Therapy (Experimental): Participants will received task specific physical therapy for 1 hour, twice a week for 6 weeks
  Interventions: Other: Task specific physical therapy

INTERVENTIONS:
Other: Task specific physical therapy — Physical Therapy based specifically on tasks that the participant os having difficulty with

SUMMARY:
The purpose of this study is to find effective physical therapy treatments for individuals who have severe multiple sclerosis. Physical therapy treatments for mild-to-moderate multiple sclerosis exists, however, very limited research has been done for physical therapy for severe multiple sclerosis (MS). In this study 10 participants diagnosed with severe MS will engage in 1-hour physical therapy sessions twice a week for 6 weeks to address limitations in standing, balancing, and bed mobility.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the feasibility, safety, and efficacy of task-specific physical therapy for persons with severe MS. The hypothesize for this study that a task-specific physical therapy program is safe, feasible, and effective in persons with severe MS.

Multiple studies have confirmed the effectiveness of task specific physical therapy for persons with MS. However,MS is a progressive disease which can lead to mild to severe disability and the studies examining the effectiveness of task specific therapy have only been conducted on persons with mild to moderate MS impairments. The small amount of research on physical therapy for persons with severe disability due to MS has only looked at the use of generalized conditioning exercises(1). Task specific therapy has been shown to be effective in persons with severe disability in non-MS neurologic disorders.(2) The effectiveness of task specific exercises on persons with severe MS not been studied. Based on the previous scientific evidence of the effectiveness of task-specific physical therapy in MS subjects with mild-to-moderate disability, there is strong scientific justification for conducting a trial of task specific therapy on persons with severe disability due to MS.

The results of this study will be presented at various conferences attended by physical therapists as well as other health care practitioners who specialize in MS care, including the American Physical Therapy Combined Sections Meeting, as well as the Consortium of Multiple Sclerosis Centers annual meeting. Additionally, upon completion of the study, we will submit a manuscript to the appropriate peer review journal.

ELIGIBILITY:
Inclusion Criteria:

1. definitive diagnosis of Multiple Sclerosis
2. Expanded Disability Status Scale (EDSS) of 7.0-8.0
3. Ability to read, understand , and sign an informed consent -

Exclusion Criteria:

1. evidence of MS exacerbation in the 4 weeks prior to starting the study
2. any orthopedic, cardiopulmonary, or non-MS neurologic symptoms that will interfere with their ability to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis Physical Frailty Functional Assessment (MSPFFA) | Will be administered twice, once at pre-intervention and once at post-intervention. The length of the intervention is 6 weeks.
  Assessment of ability to perform functional mobility tasks. The MSPFFA is a 14 item ordinal scale; the maximum score is a 56, minimom score is 14. The higher the score, the better the function and the less physically frail the person being tested is considered to be.

SECONDARY OUTCOMES:
Multiple Sclerosis Impact Scale-29 (MSIS29) | Will be administered twice, once at pre-intervention and once at post-intervention. The length of the intervention is 6 weeks.
  Self report measure of the impact of MS on the participant. The MSIS-29 is 29 item self report measure. The higher the score, the greater the impact of MS on the person person reporting bleives they have.The score is rated from 0-100 with the higher score indicating a greater impact on the individual from MS.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Karpatkin, Principal Investigator — Hunter College of City University of New York
Locations (1):
- Hunter College, Physical Therapy Department, City University of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
In addition to Individual Participant Data (IPD) the following information will be shared Study Protocol
Supporting Information: Study Protocol
Time Frame: Information to be shared will become available after publication of our findings in the appropriate peer review Journal. We expect this to happen by 12/20025 12/2025 as
Access Criteria: Access will be granted following review of the request by the PI

REFERENCES:
- [Background] Kalb R, Brown TR, Coote S, Costello K, Dalgas U, Garmon E, Giesser B, Halper J, Karpatkin H, Keller J, Ng AV, Pilutti LA, Rohrig A, Van Asch P, Zackowski K, Motl RW. Exercise and lifestyle physical activity recommendations for people with multiple sclerosis throughout the disease course. Mult Scler. 2020 Oct;26(12):1459-1469. doi: 10.1177/1352458520915629. Epub 2020 Apr 23. PMID 32323606
- [Background] Arya KN, Verma R, Garg RK, Sharma VP, Agarwal M, Aggarwal GG. Meaningful task-specific training (MTST) for stroke rehabilitation: a randomized controlled trial. Top Stroke Rehabil. 2012 May-Jun;19(3):193-211. doi: 10.1310/tsr1903-193. PMID 22668675